CLINICAL TRIAL: NCT04615611
Title: Individual beta2-adrenergic Performance Response to Salbutamol
Brief Title: Physiologic Performance Response to Salbutamol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Morten Hostrup, PhD, Associate Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: SAL-POWER
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-10

CONDITIONS: Healthy
MeSH Terms: interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- salbutamol (Experimental): salbutamol, 800 microgram from metered dose inhaler
  Interventions: Drug: salbutamol
- placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salbutamol — inhalation of salbutamol
  Arms: salbutamol
Drug: Placebo — administration of placebo
  Arms: placebo

SUMMARY:
This project aims to investigate the individual physiological response to beta2-adrenergic stimulation with salbutamol on performance-related outcomes

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years of age
* Trained individuals with maximal oxygen uptake above 55 mL/kg/min for men and 50 mL/kg/min for women
* Body mass index lower than 26

Exclusion Criteria:

* Allergy towards study drug
* Unacceptable side effects of the study drug
* Chronic disease deemed by the MD to impose a risk or severely confound the study outcomes
* Current smokers
* Use of prescription medicine
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-07 (Estimated); Primary Completion 2021-11-07 (Estimated); Study Completion 2021-11-07 (Estimated)

PRIMARY OUTCOMES:
Sprint performance | Measured ½ hour after drug administration
  Power output during maximal cycling

SECONDARY OUTCOMES:
Muscle strength | Measured ½ hour after drug administration
  Quadriceps maximal voluntary contraction
Sprint fatigue tolerance | Measured ½ hour after drug administration
  Fatigue index during maximal cycling
Cycling endurance performance | Measured ½ hour after drug administration
  4-min time trial on bike ergometer

IPD SHARING:
Plan to Share IPD: Undecided